CLINICAL TRIAL: NCT06833892
Title: H2O-F - A PROSPECTIVE, MULTI-COUNTRY, MULTI-CENTRE, MULTI-CONDITION FEASIBILITY STUDY EVALUATING THE ESTABLISHMENT OF THE NATIONAL HEALTH OUTCOMES OBSERVATORY (H2O) ECOSYSTEM
Acronym: H2O
Status: Withdrawn | Type: Observational
Why Stopped: Study was denied by Italian Ethical Committee
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Medical University of Vienna (Other); Erasmus Medical Center (Other); Charité University Hospital, Berlin, Germany (Unknown); Vall d'Hebron University Hospital, Barcelona (Unknown)
Responsible Party: Principal Investigator, Alessandra Bulotta, MD, IRCCS San Raffaele
Other Study IDs: H2O
Record Dates: First submitted 2025-02-13; First posted 2025-02-19 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: PROM

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Metastatic BC, LC, Crohn's Disease, Ulcerative Colitis or Type I and Type II Diabetes: All patients with a diagnosis of Metastatic Breast Cancer, Lung Cancer, Crohn's Disease, Ulcerative Colitis or Type I and Type II Diabetes who are treated at participating MUW centers

SUMMARY:
The primary objective of this study is to assess the progress of the national H2O Health Outcomes Observatory ecosystem towards a fully functional and operational state.

The study aims to systematically implement validated sets of PROMs (patient-reported outcomes) to enable real-time monitoring and intervention, facilitating patient-centered health care.

DETAILED DESCRIPTION:
This study is aimed to all patients with a diagnosis of Metastatic Breast Cancer, Lung Cancer, Crohn's Disease, Ulcerative Colitis or Type I and Type II Diabetes who are treated at participating MUW centers and other H2O stakeholders such as HCPs, healthcare administrators, healthcare policy makers, and academic and private sector researchers.

This is an international project that aims to systematically implement validated sets of PROMs (patient-reported outcomes) to enable real-time monitoring and intervention, facilitating patient-centered health care.

The sets of PROMs will be administered to patients during the clinical routine via online questionnaires.There are no additional procedures to the existing clinical routine.

The study includes a 6-month enrollment period and a 12-month observation period; questionnaires will be collected at baseline, 3, 6, 9, 12-month timepoints.

A total of 200 patients are expected to be enrolled among the various participating centers.

The primary objective of this study is to assess the progress of the national H2O Health Outcomes Observatory ecosystem towards a fully functional and operational state.

The secondary objectives are to

* Measure the national Health Outcomes Observatory ecosystem's usability and utility for routine care delivery and secondary research health data use cases,
* Understand stakeholders' acceptance, identify facilitators and improve and deepen the situational, contextual qualitative understanding of the perceived barriers and challenges that could prevent implementation and scalability, and
* Evaluate the infrastructure established to capture, store, and analyse integrated clinical and patient-generated health outcome data.

ELIGIBILITY:
Inclusion Criteria:

* Patients (>18 years of age) with a diagnosis of Type I or Type II Diabetes, Crohn's Disease, Ulcerative Colitis, Metastatic Breast Cancer, or Lung Cancer.
* Ability to read and understand the local language
* Participation in the H2O Registry (EK 1659/2022)
* Signed and dated informed consent form for participation in the feasibility study
* Willing and able to complete data collection using an electronic device.

Exclusion Criteria:

* Any patient who is unable or unwilling to provide explicit informed consent, or fails to meet other inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (>18 years of age) with a diagnosis of Type I or Type II Diabetes, Crohn's Disease, Ulcerative Colitis, Metastatic Breast Cancer, or Lung Cancer.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
To assess the progress of the national H2O Health Outcomes Observatory ecosystem | Data of each participant will be collected over a period of 12 months.
  The primary objective of this study is to assess the progress of the national H2O Health Outcomes Observatory ecosystem towards a fully functional and operational state using the Maturity Model

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided